CLINICAL TRIAL: NCT03662009
Title: Multi-limb Control in Parkinson's Disease: Implicit and Explicit Control of Attention
Brief Title: Multi-limb Dual-task Control in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: A.T. Still University of Health Sciences (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); University of Idaho (Other); Mayo Clinic (Other)
Responsible Party: Principal Investigator, Tara McIsaac, Professor, A.T. Still University of Health Sciences
Other Study IDs: 2017-045; 1R15NS098340-01A1 (NIH)
Record Dates: First submitted 2018-08-30; First posted 2018-09-07 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinson Disease: Observation of individuals with idiopathic Parkinson disease performing a multilimb dual task using the arm and the leg.
  Interventions: Other: multilimb dual task
- Control: Observation of healthy age-matched individuals will perform a multilimb dual task using the arm and the leg.
  Interventions: Other: multilimb dual task

INTERVENTIONS:
Other: multilimb dual task — control of arm and foot in two attentional contexts of simulated driving
  Other Names: Instructed priority; constrained accuracy

SUMMARY:
People with Parkinson disease commonly experience difficulty driving, which requires the arms and legs to do different tasks simultaneously. Driving difficulties can lead to isolation, depression, loss of independence and mobility, and increased incidence of car accidents. Through understanding the impact of Parkinson disease on mechanisms underlying attention and multi-limb control, training and rehabilitation programs can better focus on the needs of drivers with Parkinson disease. The proposed study aims to address this need by taking measures of simulated driving at one point in time. Subjects with PD are tested at a single time point when they are at their "best" point in their day and on another day when they are at their worst and are about to take their next dose of medication. Healthy age-matched subjects are not taking anti-parkinson medication so are tested at only one point.

ELIGIBILITY:
Inclusion Criteria:

* have a clinical diagnosis of mild to moderate idiopathic PD (Hoehn & Yahr stages 1-3),
* hold a valid driver's license and drive at least once a week, and
* be capable of providing informed consent and complying with study procedures. Control group participants will be healthy, neurologically intact individuals, age-matched to within 2 years of the PD subjects.

Exclusion Criteria:

* impaired global cognition (i.e., a score of < 20 on the Montreal Cognitive Assessment (MoCA) screening tool)
* sensory loss in the lower limb as assessed by clinical test of vibration perception at the ankle,
* orthopedic, visual, or neurological conditions that would prevent performance of the experimental tasks,
* inability to complete and pass the assessment testing,
* history of neurological illness such as head trauma, previous stroke, epilepsy, demyelinating disease, or
* complicating medical problems such as diabetes.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals will be recruited through collaboration with hospitals, clinics, physical therapy centers, private practice physicians and physical therapists, neurology-based fitness centers, community centers, PD support groups, online trial-matching services (e.g., FoxTrialFinder.michaeljfox.org), word of mouth, and advertising. Recruitment will be limited to the greater Phoenix metropolitan area.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Dual Task Effect on Arm and Foot Tasks | Subjects with PD: Two 90-minute sessions within a week; Healthy controls: One 90-minute session, observation of simulated driving.
  The Dual Task Effect is the performance measure of the arm and foot task, respectively, in the dual task relative to the single task, expressed as a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Tara L McIsaac, PhD, PT, Principal Investigator — A.T. Still University
Locations (1):
- A.T. Still University Arizona School of Health Sciences, Mesa, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available. Institutional infrastructure being developed.

REFERENCES:
- [Background] McIsaac TL, Benjapalakorn B. Allocation of attention and dual-task effects on upper and lower limb task performance in healthy young adults. Exp Brain Res. 2015 Sep;233(9):2607-17. doi: 10.1007/s00221-015-4333-6. Epub 2015 Jun 17. PMID 26080755
- [Background] McIsaac TL, Lamberg EM, Muratori LM. Building a framework for a dual task taxonomy. Biomed Res Int. 2015;2015:591475. doi: 10.1155/2015/591475. Epub 2015 Apr 19. PMID 25961027
- [Background] Thompson T, Poulter D, Miles C, Solmi M, Veronese N, Carvalho AF, Stubbs B, Uc EY. Driving impairment and crash risk in Parkinson disease: A systematic review and meta-analysis. Neurology. 2018 Sep 4;91(10):e906-e916. doi: 10.1212/WNL.0000000000006132. Epub 2018 Aug 3. PMID 30076275